CLINICAL TRIAL: NCT02514486
Title: Assessment of Cancer Concerns at the End of Treatment (ACE)
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 13114
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer(BC) Survivors
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Questionnaire

SUMMARY:
This study will describe patient-reported symptom burden and concerns, quality of life (QOL), and health behaviors of breast cancer(BC) survivors who have completed initial treatments (e.g., surgery, chemotherapy, and/or radiotherapy), assess the feasibility of using a web-based platform to collect patient-reported outcome (PRO) data, and evaluate provider satisfaction following delivery of an electronic health record (HER)/EPIC summary of these PROs. Secondary aims will estimate differences in referral to available services between those providers exposed to the PRO summary and historical controls. BC survivors who have completed initial treatment and present within the first year following treatment for an end of treatment (EOT)/survivorship focused visit will be the focus of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with invasive, non-metastatic BC (Stage I, II, or III) without hematogenous or distant metastases
2. Have completed initial treatment (chemotherapy, radiotherapy, and/or surgery). May still be receiving hormonal or targeted therapy (e.g., tamoxifen, aromatase inhibitors).
3. Within 1 year of completing primary treatment
4. Scheduled for an EOT visit
5. Age 18 years or older
6. Can understand written English
7. Have internet access and a working email address

Exclusion Criteria:

1. Diagnosed with non-invasive (Stage 0/DCIS) or metastatic (Stage IV) cancer or hematogenous or distant metastatic disease
2. No working email address -

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer survivors
Sampling Method: Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2014-07; Primary Completion 2018-01-19 (Actual); Study Completion 2018-01-19 (Actual)

PRIMARY OUTCOMES:
Completion of Questionnaire | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Linda Jacobs, CRNP, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States